CLINICAL TRIAL: NCT00219583
Title: A Phase 2b, Multi-Centre, Double-Blind, Placebo-Controlled, Parallel Group Dose Response Study To Assess The Efficacy and Safety Of Oral UK390,957 In Men With Premature Ejaculation
Brief Title: Assessment Of Efficacy and Safety Of UK-390,957 In Men With Premature Ejaculation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3871027
Record Dates: First submitted 2005-09-09; First posted 2005-09-22 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Ejaculation

INTERVENTIONS:
Drug: UK-390,957

SUMMARY:
Assessment of efficacy and safety UK-390,957.

ELIGIBILITY:
Inclusion Criteria:

* Premature ejaculation as defined by DSM-IV

Exclusion Criteria:

* History of erectile dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460
Dates: Start 2004-08; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy and safety

SECONDARY OUTCOMES:
Assessment of quality of sexual life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- Australia (6):
  - Pfizer Investigational Site, Bondi Junction, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Spring Hill, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Malvern, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
- Austria (2):
  - Pfizer Investigational Site, Mistelbach
  - Pfizer Investigational Site, Salzburg
- Canada (7):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, MontrÃ©al, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- Czechia (3):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Prague
- France (2):
  - Pfizer Investigational Site, Le Kremlin-Bicêtre
  - Pfizer Investigational Site, Lyon
- Germany (4):
  - Pfizer Investigational Site, Munich, Bavaria
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, München
- Israel (5):
  - Pfizer Investigational Site, Beersheba
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Jerusalem
  - Pfizer Investigational Site, Tel Aviv
  - Pfizer Investigational Site, Tel Litwinsky
- Italy (2):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Roma
- Netherlands (2):
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, The Hague
- Norway (3):
  - Pfizer Investigational Site, BodÃ¸
  - Pfizer Investigational Site, Moelv
  - Pfizer Investigational Site, Oslo
- Poland (4):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Kielce
  - Pfizer Investigational Site, Mysłowice
  - Pfizer Investigational Site, Warsaw
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
- Sweden (2):
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Balcali, Adana
  - Pfizer Investigational Site, Samanpazarı, Ankara
  - Pfizer Investigational Site, Balçova, İzmir

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3871027&StudyName=Assessment+Of+Efficacy+and+Safety+Of+UK%2D390%2C957+In+Men+With+Premature+Ejaculation++